CLINICAL TRIAL: NCT04179136
Title: The Role of Gut Microbiome on Cardiovascular Health Benefits of Dietary Lignans ( CardioFlax Study).
Brief Title: The Role of Gut Microbiome on Cardiovascular Health Benefits of Dietary Lignans (CardioFlax Study).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CardioFlax study
Record Dates: First submitted 2019-11-21; First posted 2019-11-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Cardiovascular system Polyphenols
MeSH Terms: interventions — Lignans; Linseed Oil; secoisolariciresinol

STUDY DESIGN:
Intervention Model Description: Double blinded randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High enterolactone producer's (intervention) (Active Comparator): lignan capsules contain 300 mg flaxseed (SDG) extract
  Interventions: Dietary Supplement: lignan capsules contain 300 mg flaxseed (SDG) extract
- High enterolactone producer's (Control) (Placebo Comparator): Placebo treatment matching intervention
  Interventions: Dietary Supplement: Placebo treatment matching intervention
- Low enterolactone producer's (intervention) (Active Comparator): lignan capsules contain 300 mg flaxseed (SDG) extract
  Interventions: Dietary Supplement: lignan capsules contain 300 mg flaxseed (SDG) extract
- Low enterolactone producer's (Control) (Placebo Comparator): Placebo treatment matching intervention
  Interventions: Dietary Supplement: Placebo treatment matching intervention

INTERVENTIONS:
Dietary Supplement: lignan capsules contain 300 mg flaxseed (SDG) extract — lignan capsules contain 300 mg flaxseed (SDG) extract
  Arms: High enterolactone producer's (intervention); Low enterolactone producer's (intervention)
Dietary Supplement: Placebo treatment matching intervention — Placebo treatment matching intervention
  Arms: High enterolactone producer's (Control); Low enterolactone producer's (Control)

SUMMARY:
The aim of this study is to investigate the effects of gut microbial metabolism of flaxseed lignans on cardiovascular health. Enterolactone is the main gut microbial metabolite of lignans. The study population will be stratified in low and high enterolactone producers and will investigate whether high producers will have greater benefits than low producers, and whether low producers may become high producers after daily consumption of lignans over 8 weeks. The investigators will evaluate changes in endothelial function, blood pressure, arterial stiffness, insulin resistance, lipid profile and gut microbiome composition after 8 weeks daily consumption of flaxseed lignans.

DETAILED DESCRIPTION:
Epidemiological studies have shown inverse relation between enterolactone levels and cardiovascular mortality. Participants will be stratified from first phase (NCT03573414) and then randomly allocated to treatment or placebo. Outcomes are measured at baseline and after 8 weeks post consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 20-70 years
* BMI between 18 and 35 kg/m2
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
* Are able to understand the nature of the study
* Able to give signed written informed consent
* Signed informed consent form

Exclusion Criteria:

* Medical history of cardiovascular disease including coronary artery disease, cerebrovascular disease and peripheral artery disease
* Hypertensive, as defined as SBP superior or equal to 140 mmHg, and CBP superior or equal to 90 mmHg
* Participants with BMI superior to 35 kg/m2, and BMI below 18 kg/m2
* Medical history of diabetes mellitus, metabolic syndrome, terminal renal failure or malignancies
* Abnormal heart rhythm (lower or higher than 60-100 bmp)
* Allergies to flaxseed or other significant food allergy
* Subjects under medication that can affect the cardiovascular system or on vitamin/dietary supplements.
* Subjects who have lost more than 10% of their weight in the past 6 months or are currently in a diet
* Subjects who reported participant in another study within one month before the study start
* Smoker Subjects
* Pregnant women or planning to become pregnant in the next 6 months
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in flow-mediated dilation (FMD) | Baseline vs 8 weeks post-consumption
  To investigate the effect of daily consumption of 300 mg of flaxseed (SDG) extract vs Placebo for 8 weeks on endothelium-dependent flow mediated dilation (FMD) of the brachial artery (0, 8 weeks)

SECONDARY OUTCOMES:
Change in flow-mediated dilation (FMD) | Day 0, Day1 post-consumption
  To investigate the acute effect of 300 mg of flaxseed (SDG) extract vs Placebo on endothelium-dependent flow mediated dilation (FMD) of the brachial artery after 24- hour post-consumption.
Change in office blood pressure | Day 0, Day 1 and 8 weeks post-consumption
  To investigate the effect of 300 mg flaxseed lignans (SDG) extract vs Placebo on peripheral systolic and diastolic blood pressure, and heart rate after 8 weeks daily consumption.
Change in pulse wave velocity (PWV) | Baseline vs 8 weeks post-consumption
  To determine the effect of 300 mg of lignans (SDG) vs Placebo on pulse wave velocity (PWV ) using a Sphygmocor device, after 8 weeks daily consumption
Change in augmentation Index (AIx) | Baseline vs 8 weeks post-consumption
  To determine the effect of 300 mg of lignans (SDG) vs Placebo on augmentation index (PWA) using a Sphygmocor device, after 8 weeks daily consumption
Change in Total cholesterol | Baseline vs 8 weeks post-consumption
  To investigate the effect of 300 mg Lignans (SDG) extract vs Placebo on blood lipids Total cholesterol after 8 weeks daily consumption
Change in blood inflammatory markers (IL-6) | Baseline vs 8 weeks post-consumption
  To investigate the effect of 300 mg lignans (SDG) extract vs Placebo on inflammation markers (IL-6) after 8 weeks daily consumption.
Change in glucose marker | Baseline vs 8 weeks post-consumption
  To investigate the effect of 300 mg lignans (SDG) extract vs Placebo on glucose levels (glucose) after 8 weeks daily consumption.
Change in blood lipid (HDL cholesterol ) concentrations | Baseline vs 8 weeks post-consumption
  o investigate the effect of 300 mg Lignans (SDG) extract vs Placebo on blood lipids (HDL)after 8 weeks daily consumption
Change in blood lipid (LDL cholesterol )concentrations | Baseline vs 8 weeks post-consumption
  o investigate the effect of 300 mg Lignans (SDG) extract vs Placebo on blood lipids( LDL cholesterol) after 8 weeks daily consumption
Change in blood lipid (triglycerides) concentrations | Baseline vs 8 weeks post-consumption
  o investigate the effect of 300 mg Lignans (SDG) extract vs Placebo on blood lipids (triglycerides) after 8 weeks daily consumption
Change in blood inflammatory markers (CRP) | Baseline vs 8 weeks post-consumption
  To investigate the effect of 300 mg lignans (SDG) extract vs Placebo on inflammation markers ( CRP) after 8 weeks daily consumption.
Change in insulin markers | Baseline vs 8 weeks post-consumption
  To investigate the effect of 300 mg lignans (SDG) extract vs Placebo on glucose levels (insulin) after 8 weeks daily consumption.
Change in glucose (HbA1c) markers | Baseline vs 8 weeks post-consumption
  To investigate the effect of 300 mg lignans (SDG) extract vs Placebo on glucose levels (HbA1c) after 8 weeks daily consumption.

OTHER OUTCOMES:
Change in metabolic (poly)phenol metabolite concentrations | Baseline, 24 hand 8 weeks post-consumption
  To determine the plasma levels of polyphenol metabolites after acute and chronic consumption of flaxseed lignans (SDG).Measured by liquid chromotography-mass spectrometry (LC/MS)
Change in metabolic (poly)phenol metabolite concentrations | Baseline vs 8 weeks post-consumption
  To determine the urine levels of polyphenol metabolites baseline and chronic consumption of flaxseed lignans (SDG). Measured by liquid chromotography-mass spectrometry (LC/MS)
Gut microbiome composition | Baseline vs 8 weeks post-consumption
  To investigate changes in gut microbiota composition and diversity after 8 weeks consumption of flaxseed lignans (SDG) extract.
Menopausal symptoms | Baseline vs 8 weeks post-consumption
  To investigate the effect of 300 mg flaxseed lignans (SDG) extract vs Placebo on menopausal symptoms using menopausal questionnaire for women over 45 years.
Homeostatic model assessment | Baseline vs 8 weeks post-consumption
  To assess insulin resistance (IR) using homeostatic model assessment (HOMA).

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Ana Rodriguez-Mateos, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No